# STATISTICAL ANALYSIS PLAN

# For

PROTOCOL NO.: GCAM\_TET-01

A Clinical Study of the Safety and Antibody Responses of Plasma Donors Vaccinated with a Licensed Tdap Vaccine

Protocol Version No.: 3.0 Version Date: 25Jan2021

Study Sponsor:

GCAM Inc.

## Plan Authors:

Fast-Track Drugs & Biologics, LLC 20010 Fisher Avenue, Suite G Poolesville, MD, 20837

Version Number 1.0

Date: 08Nov2021

# STATISTICAL ANALYSIS PLAN PROTOCOL NO.: GCAM-TET-01

A Clinical Study of the Safety and Antibody Responses of Plasma Donors Vaccinated with a Licensed Tdap Vaccine

Date: 08 November 2021

| Prepared by: | Date: |
|--------------|-------|
| Reviewed by: | Date: |
| Reviewed by: | Date: |

Statistical Analysis Plan Protocol GCAM-TET-01 Version 1.0
Date: 08Nov2021

# **Table of Contents**

| 1. | List of Abbreviations | 4 |
|---|---|---|
| 2. | Introduction | 5 |
| 3. | Protocol Summary 3.1. Study Objectives 3.2. Study Design 3.3. Study Endpoints | 6<br>6 |
| 4. | Definition of Analysis Sets | 9 |
| 5. | Assessment and Justification of Study Endpoints 5.1. Safety Endpoints 5.2. Efficacy Endpoints 5.3. Baseline and other Assessments | 9<br>11 |
| 6. | Hypotheses to be Tested | 12 |
| 7. | Sample Size | 12 |
| 8. | Data Quality Assurance | 12 |
| 9. | Statistical Considerations 9.1. General Considerations 9.2. Participant Accountability and Protocol Deviations 9.3. Demographics, Pre-donation Screening, and Treatment Compliance 9.4. Immunizations, Prior and Concomitant Medications 9.5. Analysis of Safety Endpoints 9.6. Clinical Laboratory Data 9.7. Analysis of Efficacy Endpoints | 12<br>13<br>13<br>13 |
| 10. | Handling of Missing Data and Missing Date | 15 |
| 11. | Validation of Programming Code. | 15 |
| 12. | Changes to Planned Analyses | 15 |
| 13. | Appendix A: Table and Figure Shells | 16 |
| 14. | Appendix B: Listing Shells | 36 |

# 1. List of Abbreviations

| Abbreviation | Definition |
|--------------|--------------------------------------------------------|
| AE | Adverse event |
| CRF | Case report form |
| CSR | Clinical Study Report |
| ELISA | Enzyme-linked immunosorbent assay |
| I/E | Inclusion/Exclusion |
| HAV | Hepatitis A virus |
| HBsAg | Hepatitis B surface antigen |
| HBV | Hepatitis B virus |
| HCV | Hepatitis C virus |
| HIV | Human Immunodeficiency Virus |
| IU/mL | International Unit/ Mililiter |
| ITT | Intent-to-treat |
| MedDRA | Medical Dictionary for Regulatory Activities |
| max | Maximum |
| min | Minimum |
| msec | Milliseconds |
| n | Number of observations |
| PI | Principal Investigator |
| PP | Per-protocol |
| QA | Quality Assurance |
| RPR | Rapid plasma reagin |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SOC | System, Organ, Class |
| SOP | Standard operating procedure |
| Tdap | Tetanus toxoid, diphtheria toxoid, acellular pertussis |
| US | United States |
| WHO | World Health Organization |

#### 2. Introduction

This analysis plan describes the core set of table summaries, data listings, graphic representations, and pre-planned statistical analyses to address the study objectives for protocol number GCAM-TET-01. In addition, *post hoc* exploratory analyses may also be performed to aid in interpretation of the data. Any prospective changes to the plan will be made, reviewed, and approved before the database is locked. Changes to the planned conduct of the analysis will be documented and justified in Clinical Study Report (CSR).

This SAP describes Safety evaluations, based on clinical parameters, laboratory testing and assessment of adverse events (AEs) etc., and efficacy evaluations based on anti-tetanus anitibody titers levels.

# 3. Protocol Summary

# 3.1. Study Objectives

# Primary Objective

 To assess the safety of a licensed Tdap vaccine when given every 3 months for a total of 5 immunizations over a period of 12 months.

# Secondary Objectives

 To assess anti-tetanus antibody titers over time of a licensed Tdap vaccine when given every 3 months for a total of 5 immunizations over a period of 12 months and for 6 months after the final immunization.

# 3.2. Study Design

This is a prospective, open label, single-arm, multi-center, Phase 2 study measuring the safety and tetanus antibody responses to Tdap vaccine administered to plasma donors every 3 months ±1 week for 12 months (5 vaccinations) with a 6 month follow-up after the last vaccination. After obtaining informed consent and screening for eligibility including plasmapheresis donor eligibility, subjects will have other baseline assessments performed and if eligible, will receive the scheduled vaccinations, will be assessed for adverse events (AEs) and have plasma samples collected with antibody titers reported each month thereafter for 11 months, and then at 1 and 6 months after the last vaccination. Subjects will undergo plasmapheresis prior to the second through the fifth vaccination and at the 1 month and 6 month post vaccination follow-up visits. As these subjects are participating in a standard donor plasmapheresis donor program, assessments for donor eligibility and routine plasmapheresis will be performed; however, only the data specifically required to meet the objectives of this study will be collected.

The study time and events schedule is shown in <u>Table A</u>. In addition to these study specific assessments routine screening procedures to assure plasma donor suitability was also performed. Some of the routine procedures performed as part of plasma donor screening evaluations such as vital signs, physical examinations, or laboratory tests were reported as AEs (if appropriate) on an AE eCRF.

## 3.3. Study Endpoints

#### Safety Endpoints:

 Incidence, severity, and relationship of AEs to the study vaccine in the time period between vaccinations and for the overall study period.

#### Efficacy endpoints:

- Anti-tetanus antibody titer levels after each vaccination presented at geometric means (GeoMean) over time.
- The numbers and percentages of subjects whose post vaccination antibody levels are
   1U/mL; ≥5 IU/mL to 10 IU/mL; > 10 IU/mL to 15 IU/mL; and > 15 IU/mL after each vaccination.

Table A: Time and Events Schedule

| Study Phase | Screening | | | | | Vi | sits (Mo | onth 0 to | Month | 12 ± 1 v | week) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Month | -7 to -1 | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 |
| | days | | | | | | | | | | | | | |
| Visit Number | 1 | 2/3 | 4 | 5 | 6/7 | 8 | 9 | 10/11 | 12 | 13 | 14/15 | 16 | 17 | 18/19 |
| Study Specific Proced | lures for whic | h dat | a are | recor | rded o | n an eC | RF | | | | | | | |
| Consent | X | | | | | | | | | | | | | |
| Eligibility checklist <sup>a</sup> | X | X | | | X | | | X | | | X | | | X |
| Demographics | X | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | |
| Medications | X | X | | | X | | | X | | | X | | | X |
| Vaccination | | 1 | | | 2 | | | 3 | | | 4 | | | 5 |
| AEs | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Plasma sample for | X | | X | X | X | X | X | X | X | X | X | X | X | X |
| anti-tetanus and anti- | | | | | | | | | | | | | | |
| diphtheria antibody | | | | | | | | | | | | | | |
| titer <sup>b</sup> | | | | | | | | | | | | | | |
| Urinalysis/ serum | | X | | | X | | | X | | | X | | | X |
| creatinine <sup>c</sup> | | | | | | | | | | | | | | |
| Diary card review <sup>d</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Procedures performe | d as part of re | outine | e plas | ma d | onor te | esting ar | nd pher | esis | | | | | | |
| Medical history <sup>e</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Body weight | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Infectious diseases <sup>f</sup> | X | | | | | | | | | | | | | |
| Immunization record | X | | | | | | | | | | | | | |
| Medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Pre-donation | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| screening | | | | | | | | | | | | | | |
| examination <sup>g</sup> | | | | | | | | | | | | | | |
| Plasmapheresis | | | P | lasma | donati | ons may | occur 2 | | | | least one- | calendar | day be | ween |
| | | | | | | | | de | onations | 3. | | | | |

Statistical Analysis Plan Protocol GCAM-TET-01 Version 1.0 Date: 08Nov2021 <sup>a</sup>At screening, the reasons a subject is not eligible for the study (screen failure) will be captured on a Reasons Not Eligible eCRF. Subjects will be checked to ensure that they meet study eligibility criteria prior to each vaccination. If not eligible, a Reasons not Eligible for Vaccination eCRF will be completed.

<sup>b</sup>Tetanus and diphtheria antibody test samples will be collected, frozen and tested at a later date. Samples are collected from plasma donations performed at these visits. If a plasmapheresis was not scheduled or performed at this visit (± 1 week) then a blood sample collected for plasma separation may be used instead.

<sup>c</sup>Serum creatinine and urinalysis - measured 1-3 days after each study vaccination. If the subject does not return to the center within this time frame, the sample should be collected and tested at the next visit to the center.

<sup>d</sup>The subject's diary card will be reviewed at each monthly visit for recording of AEs and medications.

eMedical history is updated at all visits after the screening visit including reports of pregnancy by female participants.

<sup>f</sup>Anti-HIV-1/2, HBsAg, Anti-HCV, SPE/RPR, Indirect Coombs, and PCR testing for HIV-1, HBV and HCV, HAV, Parvovirus B19 are tested from plasma samples collected from two sequential plasma donations and must be negative for a subject to be eligible for the study. Infectious disease testing is also performed on plasma samples collected from plasma donations and if a subject is positive for any of these infectious diseases, they will be taken off study. In addition, RPR (syphilis test) is performed every 4 months.

<sup>g</sup>Pre-donation screening assessments include a full physical exam performed annually, vital signs and hematocrit and total protein at each donation. If the subject is already a donor of record, the full physical examination will only be performed when regularly scheduled

Table A Continued: Time and Events Schedule

| | Follow-Up 1 | Follow-Up 2 |
|---|---|---|
| Month | 13 | 18 |
| Visit Number | 20 | 21 |
| Medications | X | X |
| AEs | X | X |
| Plasma sample for anti-tetanus and anti-diphtheria antibody titer | X | X |
| Diary card review | X | X |
| Subject disposition | | X |
| Medical history | X | X |
| Body weight | X | X |
| Medications | X | X |
| Pre-donation screening examination | X | X |
| Subject Disposition <sup>a</sup> | | X |

<sup>&</sup>lt;sup>a</sup> The final disposition of the subject will be reported on a Subject Disposition eCRF including if the subject completed the full study or withdrew early and the reason for early withdrawal. This eCRF will be completed at an earlier visit if the subject withdrew from the study.

8

.0

## 4. Definition of Analysis Sets

**Intention-to-treat (ITT) Population:** The ITT population will consist of all subjects who are enrolled into the study and received any amount of investigational product. This population will be used in safety analysis.

**Per-protocol (PP) Population:** The per-protocol population will consist of all subjects in the ITT population who received all 5 TdaP vaccinations and completed the 6 month follow-up visit after the final vaccination.

# 5. Assessments and Justification of Study Endpoints

The schedule of Assessments for the study is shown in **Table A**.

# 5.1. Safety Endpoints

**Adverse Events:** AEs will include any treatment emergent unfavorable and unintended sign or symptom inleuding abnormal laboratory findings that occur at any time after the subject has signed informed consent until the second follow up visit after the last study vaccination, whether or not considered drug related.

<u>Severity:</u> All AEs will be assessed for severity by the investigator. Assignment of grade based on the intensity of symptoms and the degree of limitation of usual daily activities will be done according to severity using the following criteria:

**Mild:** The AE did not cause interference with the subject's activity.

**Moderate:** The AE produced limited functional impairment and may have required therapeutic intervention. The AE produced no sequelae.

**Severe:** The AE resulted in significant impairment of function and may have lead to temporary inability to resume the subject's normal life pattern.

**Relationship:** The degree of certainty for which the AE/SAE is attributed to the investigational product or alternative causes will be determined by the investigator's use of clinical judgment in conjunction with the assessment of a plausible biologic mechanism, a temporal relationship between the onset of the event in relation to receipt of the investigational product, and identification of possible alternate etiologies including underlying disease, concurrent illness or concomitant medications. Only a physician can make this determination.

The following drug relationships will be used for this clinical study:

**Unrelated:** There is no temporal relationship between the event and the administration of the product or the event is clearly due to the subject's medical condition, other therapies, or accident.

**Unlikely:** There is evidence of exposure to the product but there is another more likely cause of the event.

**Possible:** There is some temporal relationship between the event and the administration of the product and the event is unlikely to be explained by the subject's medical condition or other therapies.

**Probable:** The temporal relationship between the event and the administration of the product is compelling, and the subject's medical condition and other therapies cannot explain the event.

**Definite:** The event follows a reasonable temporal sequence from administration of the medication or follows a known or suspected response pattern to the medication.

The categories of definite, probable, and possible will be considered investigational product related with regards to summary statistics.

<u>AE Actions and Outcomes:</u> For each AE that is reported the actions taken with respect to study drug including: 1) none, 2) study drug discontinued, or 3) study drug interrupted will be recorded on the AE CRF. Also, outcomes will also be recorded including: 1) Fatal; 2) Resolved without sequelae; 3) Resolved with sequelae; 4) Ongoing, and 5) Unknown. If the AE required any treatment, this will also be recorded.

<u>Serious Adverse Events (SAE)</u>: An AE or suspected adverse reaction is considered "serious" if, in the view of either the PI or Sponsor, it results in any of the following outcomes:

- Death
- Life-threatening adverse event
- Inpatient hospitalization or prolongation of existing hospitalization
- Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Is an important medical event that may not result in death, be life threatening, or require hospitalization, but based on appropriate medical judgment may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed above.

<u>Solicited Adverse Events:</u> Solicited AEs will be those AEs that occur for up to 3 days after each vaccination. The severity rating scale in <u>Table B</u> will be provided to the subject, to assess the severity of solicited AEs recorded in the diary. At the diary review, if any items are checked, a clinician will review these with the subject to confirm that the appropriate severity rating was selected.

Table B: Severity Rating Scale for Solicited Adverse Events

| Adverse Event | Grade 0 | Grade 1 | Grade 2 | Grade 3 |
|---|---|---|---|---|
| Injection site redness | None | 2.5 – 5 cm | 5.1 – 10 cm | > 10 cm |
| Urticaria or other rash | None | No interference with activity | Some interference with activity | Significant; prevents daily activity |
| Injection site<br>tenderness/ pain | None | No interference with activity | Some interference with activity | Significant; prevents daily activity |

10

| Adverse Event | Grade 0 | Grade 1 | Grade 2 | Grade 3 |
|---|---|---|---|---|
| Injection site<br>swelling | None | 2.5 – 5 cm and does<br>not interfere with<br>activity | 5.1 – 10 cm or interferes<br>with activity | > 10 cm or prevents<br>daily activity |
| Fever | None | 100.4 - 101.1 | 101.2 - 102.0 | 102.1 – 104 |
| Headache | None | No interference with activity | Repeated use of<br>nonnarcotic pain reliever ><br>24 hours or some<br>interference with activity | Significant; any use<br>of narcotic pain<br>reliever or prevents<br>daily activity |
| Nausea/vomiting | None | No interference with activity or 1 – 2 episodes/24 hours | Some interference with activity or > 2 episodes/24 hours | Prevents daily<br>activity, requires<br>outpatient IV<br>hydration |
| Chills, fatigue, joint<br>pain malaise, muscle<br>weakness (myalgia) | None | No interference with activity | Some interference with activity | Significant; prevents daily activity |

# 5.2. Efficacy Endpoints

When plasmapheresis is scheduled during one of the clinical protocol monthly study visits, a sample of the plasma collected during plasmapheresis will be collected. Samples will be stored at ≤ -20°C until tested and will be tested throughout the study shortly after collection. Tetanus antibody responses will be measured at a central laboratory using an enzyme-linked immunosorbent assay (ELISA) [VaccZyme Tetanus Toxoid IgG − Binding Site] and expressed as international units per mL (IU/mL).

#### 5.3. Baseline and Other Assessments

A complete medical history and demography (gender, age, race, and ethnicity) will be collected at the screening visit. Medications being taken by the subject in the 7-day period prior to the first vaccination through the completion of the study along with complete immunization history will be recorded and reported on an eCRF.

Vitals signs, full physical examinations and hematocrit and total protein determinations as part of the routine plasmapheresis will be assessed during pre-donation screening.

Infectious disease testing will be performed on all plasma samples collected from plasma donations and if a subject is positive for any of these infectious diseases, they will be taken off study. In addition, RPR (syphilis test) is performed every 4 months. If the subject is a first time donor, they must have two sequential plasma donations that are negative for the following infectious diseases to be eligible for plasmapheresis: Anti-HIV-1/2, HBsAg, Anti-HCV, SPE/RPR, Indirect Coombs, and PCR testing for HIV-1, HBV and HCV, HAV, and Parvovirus B19.

An eligibility checklist will be completed at screening. If the subject is not eligible for the study, a Reasons Not Eligible eCRF will be completed.

A dipstick urinalysis will be performed that tests for protein, blood, leukocyte esterase, nitrates, pH, specific gravity, ketones, bilirubin, and glucose. A blood sample will also be collected for a serum creatinine test. These tests will be performed to monitor for the possible development of immune complex-mediated glomerular disease.

Anti-diphtheria antibody levels will be measured at a central laboratory using the EUROIMMUN Anti-Diphtheria Toxoid ELISA (IgG). High anti-diphtheria titers will be assessed for an association with an increase in reactogenicity.

# Hypotheses to be Tested

Hypothesis tests will be performed in order to determine if there is an association between reactogenicity and anti-diphtheria titers. Null Hypothesis of no association between reactogenicity and anti-diphtheria titers will be tested on Slope obtained using simple linear regression analysis at alpha=0.01 using two-sided tests.

# 7. Sample Size

One hundred subjects will be enrolled in this study.

# 8. Data Quality Assurance

Data quality is maintained by ensuring accuracy of data, reviewing protocol prior to study start, auditing data according to GCP and periodic site monitoring by sponsor's designees. Written instructions will be provided for collection, preparation, and shipment of blood spot samples.

The Sponsor's designees will review source documents for accuracy and completeness during on-site and remote monitoring visits and any discrepancies will be resolved with the PI, as appropriate.

Significant and/or repeated noncompliance will be investigated and remedial action instituted when appropriate. Failure to comply with remedial actions may result in study site termination and regulatory authority notification.

#### 9. Statistical Considerations

## 9.1. General Considerations

Descriptive statistics will be used to present study data. Continuous variables will be presented as number of observations (n), mean, standard deviation (SD), median, minimum (min) and maximum (max) values. Categorical and dichotomous variables will be presented as counts and percentages. As it is expected that titers will not be normally distributed, geometric means (GeoMean) will be used to summarize anti-tetanus and anti-diphtheria antibody titers. All data will be presented in listings.

Analyses will be done using SAS v9.4.

12

# 9.2. Participant Accountability and Protocol Deviations

The disposition of all study subjects will be summarized including the total numbers screened, eligible, enrolled, ITT, per-protocol, withdrawn, and completed. Accountability data including study termination and reason will be provided in a summary table and listing for all subjects who were enrolled. A listing of all protocol deviations will be provided.

## 9.3. Demographics, Pre-donation Screening and Treatment Compliance

Subject demographics which includs age (years), gender, ethnicity and race will be summarized for the ITT and Per-protocol population. Pre-donation screening for plasmapheresis check includes full physical examinations, vital signs, total proteins and hematocrit at each donation, will be summarized by visit and listed by subject and visit. Compliance with scheduled vaccinations will also be summarized, including number of doses and total dose of investigational product. Protocol compliance will be presented as percentages of subjects attending scheduled visits over the duration of the study.

## 9.4. Immunizations, Prior and Concomitant Medications

Prior and comcomitant medications will be listed by subject. Medications and treatments with an end date prior to the first dose of study drug will be considered prior medications and will be noted in listing. If the date is partial or unknown, then medication will be considered as concomitant. Any prior immunizations will be listed by subject.

# 9.5. Analysis of Safety Endpoints

Treatment emergence will be evaluated for all AEs. Treatment-emergent adverse events (TEAEs) are those that occur on or after the same date and time of first dose of study drug. TEAEs will be coded using the most recent version of the Medical Dictionary of Regulatory Affairs (MedDRA) by assigning a preferred term and will be grouped by system, organ, and class (SOC) designation. AEs occurring after each vaccination up to the time of the next vaccination and separately over the whole study period will be summarized. Separate tables will be provided for solicited AEs reported within the 3 day period after each vaccination.

Each AE will be counted once only by preferred term for a given study subject within each post vaccination time period prior to the next vaccination or up to the 6-month follow-up visit after the last vaccination. If the same AE occurred on multiple occasions, the highest severity and relationship to investigational product will be assumed within each time period.

The summary tables will include an overall summary of number and percentage of subjects reporting each TEAE, summary by relationship, summary by severity will be presented by each vaccination period and overall.

Listings of each individual AE including start date, stop date, severity, relationship, duration, outcome, and actions taken will be provided.

Reactogenicity is defined as the total count of a set of solicited AEs that are expected after a vaccine. A regression analysis will be performed with reactogenicity as the dependent variable and anti-diphtheria titers as the independent variable to determine if there is an association. Anti-diphtheria titer is not expected to be normally distributed and will be natural log transformed. Null Hypothesis of no association between reactogenicity and anti-diphtheria titers will be tested on

Slope obtained using simple linear regression analysis at alpha=0.01 using two-sided tests. The null hypothesis states that the slope is equal to zero, and the alternative hypothesis states that the slope is not equal to zero. No adjustment for covaiates will be made. The following SAS procedure PROC REG may be used.

```
Proc reg data=data;
Model reactogenicity =log(anti_diptheria_titers);
Run:
```

In addition, 2x2 tables will be created with presence or absence of moderate to severe reactogenicity versus high or not anti-diphtheria titers. Cut points of 75<sup>th</sup> percentile or 90<sup>th</sup> percentile of the anti-diphtheria titers will be used to define high level. The following SAS procedure PROC FREQ may be used.

```
Proc freq data=data;
Table reactogenicity*anti_diptheria_titers/ nopercent nocol;
Weight count;
Run:
```

# 9.6. Clinical Laboratory Data

Laboratory data for urinalysis results and serum creatinine levels will be presented as summary statistics by visit as well as in by-subject data listings. The number and percentage of subjects with serum creatinine > 1.5 x upper limit of normal and urine indicative for proteinuria (2+) or hematuria (blood  $\geq$  50 erythrocytes/ $\mu$ L).

# 9.7. Analysis of Efficacy Endpoints

Tetanus antibody titers (IU/mL) will be presented as geometric mean (GeoMean), minimum and maximum concentrations after each vaccination at all collection time points. Linear plots of the geometric mean ± Standard errors of Tetanus antibody titers will be provided by each collection time points.

The numbers and percentages of subjects whose post vaccination anti-tetanus antibody levels are <5 IU/mL; ≥5 IU/mL to 10 IU/mL; >10 IU/mL to 15 IU/mL; and, >15 IU/mL will be presented in a table over time. The percentages of subjects in each of these categories will also be presented in scatter plot over collection time.

14

# 10. Handling of Missing Data and Missing Date

Missing Data will not be imputed.

Missing dates are handled as follows:

- Missing day: The first day of the month will be used.
- Missing Month: The first month of the year will be used.
- Completely missing dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.

# 11. Validation of Programming Code

All SAS code used to generate tables, listings, and figures will be validated and reviewed before being finalized. The validation process will be used to determine that the numbers are produced by a statistically valid method and that the execution of the computations is correct. Qualified personnel who have not previously been involved in the production of the original programming code will perform the validation procedures. Methods of validation include independent programming and comparison to data listings. Tables will be reviewed for accuracy, consistency with this plan, consistency within tables, and consistency with corresponding output. Once validation is complete, a quality control reviewer will perform a final review of the documents for accuracy and consistency. Upon completion of validation and quality review procedures, all documentation will be collected and filed in the study documentation files at Fast-Track.

# 12. Changes to Planned Analyses

There are no changes between protocol-defined statistical analyses and those presented in this SAP.

15

# 13. Appendix A: Table and Figure Shells List of Tables and Figures

| Table 1: | Summary of Subject Disposition - All Consented Subjects | 17 |
|---|---|---|
| Table 2: | Reasons for Not Meeting Eligibility Criterion - Not Enrolled Subjects | 18 |
| Table 3: | Demographics and Subject Characteristics | 19 |
| Table 4: | Summary of Protocol and Treatment Compliance | 20 |
| Table 5: | Summary of Plasmapheresis Check by Visit | 21 |
| Table 6: | Summary of Treatment-emergent Adverse Events – ITT Population | 22 |
| Table 7: | Summary of Solicited Treatment-emergent Adverse Events – ITT Population | 23 |
| Table 8: | Summary of Treatment-emergent Adverse Events by System Organ Class and Preferem – ITT Population | |
| Table 9: | Summary of Solicitedd Treatment-emergent Adverse Events by System Organ Class<br>Preferred Term – ITT Population | |
| Table 10: | Summary of Subjects with Treatment-emergent Adverse Events by Severity and Relationship - ITT Population | 26 |
| Table 11: | Contingency Table of Table of Reactogenicity and Anti-diptheria titers - ITT Popula | tion 27 |
| Table 12: | Summary of Serum Creatinine and Urinalysis Tests – ITT Population | 28 |
| Table 13: | Summary of Anti-tetanus Antibody Titers (IU/mL). | 29 |
| Table 14: | Summary of Anti-diphtheria Antibody Titers (IU/mL) | 30 |
| Table 15: | Number (%) of Subjects with Post Vaccination Anti-tetanus Antibody Levels | 31 |
| Figure 1: | Regression Plot of Reactogenicity versus Anti-diptheria titers - ITT Population | 32 |
| Figure 2: | Plot of GeoMean (± SD) of Tetanus Antibody Titers | 33 |
| Figure 3: | Scatter Plot of Percentage of Subjects with Post Vaccination Anti-tetanus Antibody l - ITT Population | |
| Figure 4: | Scatter Plot of Percentage of Subjects with Post Vaccination Anti-tetanus Antibody l - Per-protocol Population | |

Table 1: Summary of Subject Disposition - All Consented Subjects

| Disposition Category | Total |
|---------------------------------------------------------|----------|
| Total Consented | XX |
| Total Eligible | xx |
| Enrolled and Received First Vaccination | xx |
| Data below is n (%) of enrolled | |
| Intention-to-treat (ITT) Population | xx (x.x) |
| Per-protocol (PP) Population | xx (x.x) |
| Subjects completing study (Completed Month 18 visit) | xx (x.x) |
| Subjects terminating early <sup>a</sup> | |
| AE or SAE | xx (x.x) |
| Protocol violation | xx (x.x) |
| Subject did not comply with protocol | xx (x.x) |
| Continued participation will pose a risk to the subject | xx (x.x) |
| Pregnancy | xx (x.x) |
| Subject withdrew participation | xx (x.x) |
| Subject no longer eligible for study participation | xx (x.x) |
| Other | xx (x.x) |

<sup>&</sup>lt;sup>a</sup>Subjects may have been terminated for more than one reason, thus numbers will not add up to the total numbers of subjects.

17

<sup>&</sup>lt;Program Name: Time and Date>

Table 2: Reasons for Not Meeting Eligibility Criterion - Not Enrolled Subjects

| Reason | n= xx |
|----------------------------|-----------|
| Informed consent Withdrawn | xx (x.x%) |
| (List all reasons) | xx (x.x%) |

Table 3: Demographics and Subject Characteristics

| Characteristic | ITT | Per-protocol |
|-------------------------------------------|-------------|--------------|
| | N=xx | N=xx |
| Gender | | |
| Male | xx (x.x%) | xx (x.x%) |
| Female | xx (x.x%) | xx (x.x%) |
| Age (years at date of consent) | | |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) |
| Median | xx.x | XX.X |
| Min-Max | (xx - xx) | (xx - xx) |
| Maximum | | |
| Race | | |
| Black or African American | xx (x.x%) | xx (x.x%) |
| American Indian or Alaskan Native | xx (x.x%) | xx (x.x%) |
| Asian | xx (x.x%) | xx (x.x%) |
| Native Hawaiian or Other Pacific Islander | xx (x.x%) | xx (x.x%) |
| White | xx (x.x%) | xx (x.x%) |
| OtherUnknown | xx (x.x%) | xx (x.x%) |
| | xx (x.x%) | xx (x.x%) |
| Ethnicity | | |
| Hispanic or Latino | xx (x.x%) | xx (x.x%) |
| Not Hispanic or Latino | xx (x.x%) | xx (x.x%) |
| Not Reported | xx (x.x%) | xx (x.x%) |

Table 4: Summary of Protocol and Treatment Compliance

| | ITT |
|---------------------------------------|-------------|
| | N=xx |
| Protocol compliance rate <sup>a</sup> | |
| Month 0 | xx.x% |
| Month 3 | xx.x% |
| Month 6 | xx.x% |
| Month 9 | xx.x% |
| Month 12 | xx.x% |
| Number of Tdap vaccinations | |
| Mean (SD) | xx.x (x.xx) |
| Median | XX.X |
| Min-Max | (xx - xx) |
| Total Tdap vaccination dose (mL) | |
| Mean (SD) | xx.x (x.xx) |
| Median | XX.X |
| Min-Max | (xx - xx) |

<sup>&</sup>lt;sup>a</sup>Protocol compliance is presented as percentages of subjects attending each scheduled treatment visit.

<sup>&</sup>lt;Program Name: Time and Date>

Table 5: Summary of Plasmapheresis Check by Visit - ITT Population

| Visit | | n (%) |
|---|---|---|
| Screening | Eligible for Plasmapheresis | |
| | Yes | xx.x (x.xx) |
| | No, Temporary | xx.x (x.xx) |
| | No, Permanent | xx.x (x.xx) |
| | If "No, Temporary", Inclusion Criteria not Met | |
| | Temperature: 97.0 - 99.5 °F | xx.x (x.xx) |
| | Blood Pressure: 90 - 180/50 - 90 mmHg | xx.x (x.xx) |
| | Pulse: 50 - 100 beats/min | xx.x (x.xx) |
| | (List all criteria not met) | |
| (Repeat for all visits) | | |

Table 6: Summary of Treatment-emergent Adverse Events - ITT Population

| | Vaccination Number | | | | | |
|---|---|---|---|---|---|---|
| | 1<br>N=xx | 2<br>N=xx | 3<br>N=xx | 4<br>N=xx | 5<br>N=xx | Overall<br>N=xx |
| Number of AEs | XX | xx | XX | XX | xx | xx |
| Number of SAEs | xx | XX | XX | XX | XX | XX |
| Number of AEs related to study product | xx | XX | XX | XX | XX | xx |
| Number (%) of subjects with | | | | | | |
| At least one AE | xx (x.x%) | xx (x.x%) | xx (x.x%) | xx (x.x%) | xx (x.x%) | xx (x.x%) |
| At least one SAE | xx (x.x%) | xx (x.x%) | xx (x.x%) | xx (x.x%) | xx (x.x%) | xx (x.x%) |
| At least one AE related to study product | xx (x.x%) | xx (x.x%) | xx (x.x%) | xx (x.x%) | xx (x.x%) | xx (x.x%) |
| Number of AEs by severity | | | | | | |
| Mild | xx | XX | XX | XX | XX | XX |
| Moderate | xx | xx | XX | XX | xx | XX |
| Severe | xx | xx | XX | xx | xx | xx |
| Number of AEs by relationship to study | | | | | | |
| product | xx | xx | XX | XX | xx | XX |
| Unrelated | xx | xx | XX | XX | xx | XX |
| Unlikely | xx | xx | XX | XX | xx | XX |
| Possible | xx | xx | xx | xx | xx | XX |
| Probable | xx | xx | XX | XX | xx | XX |
| Definite | | | | | | |
| Serious? | xx | xx | XX | xx | xx | xx |
| Yes | xx | XX | XX | XX | XX | XX |
| No | | | | | | |

Note: AEs occurring after each vaccination up to the time of the next vaccination is summarized.

<sup>&</sup>lt;Program Name: Time and Date>

Table 7: Summary of Solicited Treatment-emergent Adverse Events - ITT Population

| | Vaccination Number | | | | | |
|---|---|---|---|---|---|---|
| | 1<br>N=xx | 2<br>N=xx | 3<br>N=xx | 4<br>N=xx | 5<br>N=xx | Overall<br>N=xx |
| Number of Solicited TEAEs | XX | XX | XX | XX | XX | XX |
| Number of AEs related to study product | XX | xx | XX | XX | XX | XX |
| Number (%) of subjects with | | | | | | |
| At least one soliciated TEAE | xx (x.x%) | xx (x.x%) | xx (x.x%) | xx (x.x%) | xx (x.x%) | xx (x.x%) |
| At least one AE related to study product | xx (x.x%) | xx (x.x%) | xx (x.x%) | xx (x.x%) | xx (x.x%) | xx (x.x%) |
| Number of Solicited TEAEs by severity | | | | | | |
| Mild | xx | xx | xx | XX | xx | XX |
| Moderate | xx | xx | XX | XX | XX | XX |
| Severe | xx | XX | XX | XX | XX | XX |
| Number of Solicited TEAEs by | | | | | | |
| relationship to study product | xx | xx | XX | XX | XX | XX |
| Unrelated | xx | xx | XX | XX | XX | XX |
| Unlikely | xx | xx | XX | XX | xx | XX |
| Possible | xx | xx | XX | XX | XX | XX |
| Probable | xx | xx | XX | XX | XX | XX |
| Definite | | | | | | |

Note: Solicited AEs reported within the 3 day period after each vaccination is summarized.

N = Number of Subjects

<sup>&</sup>lt;Program Name: Time and Date>

Table 8: Number (%) of Subjects with Treatment-emergent Adverse Events by System Organ Class and Preferred Term - ITT Population

| | Vaccination Number | | | | | |
|---|---|---|---|---|---|---|
| | 1 | 2 | 3 | 4 | 5 | Overall |
| System, Organ, Class/ | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx |
| Preferred Term | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| SOC 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: Subjects are counted only once within each system organ class and preferred term.

<sup>&</sup>lt;Program Name: Time and Date>

Table 9: Number (%) of Subjects with Solicited Treatment-emergent Adverse Events by System Organ Class and Preferred Term - ITT Population

| | Vaccination Number | | | | | |
|---|---|---|---|---|---|---|
| | 1 | 2 | 3 | 4 | 5 | Overall |
| System, Organ, Class/ | N=xx | N=xx | N=xx | N=xx | N=xx | N=xx |
| Preferred Term | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| SOC 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SOC 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>:</sup> Note: Solicited AEs reported within the 3 day period after each vaccination is summarized.

Subjects are counted only once within each system organ class and preferred term.

<sup>&</sup>lt;Program Name: Time and Date>

Table 10: Summary of Subjects with Treatment-emergent Adverse Events by Severity and Relationship - ITT Population

| | Number of Subjects (%) (N=xx) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| System, Organ, Class\<br>Preferred Term | Mild Mo | | Mod | Ioderate Sev | | ere | All Gi | All Grades | |
| | R | NR | R | NR | R | NR | R | NR | R + NR |
| SOC<br>Preferred Term | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: Subjects are counted only once by preferred term at the highest severity grade and closest relationship to the investigational product. R= Related to investigational product (possible, probable, definite). NR = Not related to investigational product (unrelated, unlikely).

Table 11: Contingency Table of Reactogenicity and Anti-diptheria titers - ITT Population

| Vaccination | Moderate to Severe | Anti-dipthe | eria Titers | |
|-------------|--------------------|-------------|-------------|-----------|
| Number | Reactogenicity | High = Yes | High = No | Total |
| | | n (%) | n (%) | n (%) |
| 1 | Present | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Absent | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Total | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | Present | xx (xx.x) | xx (xx.x) | AA (AA.A) |
| | Absent | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Total | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | Present | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Absent | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Total | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 | Present | xx (xx.x) | xx (xx.x) | AA (AA,A) |
| | Absent | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Total | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 5 | Present | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Absent | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Total | xx (xx.x) | xx (xx.x) | aa (aaia) |
| Overall | Present | xx (xx.x) | xx (xx.x) | |
| | Absent | xx (xx.x) | xx (xx.x) | |
| | Total | xx (xx.x) | xx (xx.x) | |

Note: Reactogenicity is defined as the total count of a set of solicited AEs that are expected for up to 3 days after each vaccination. Cut points of 75<sup>th</sup> percentile of the anti-diphtheria titers is used to define high level. < Program Name: Time and Date >

Table 12: Summary of Serum Creatinine and Urinalysis Tests - ITT Population

| Parameter (Unit) | | Month 0 | Month 3 | Month 6 | Month 9 | Month 12 |
|---|---|---|---|---|---|---|
| | | n (%) | n (%) | n (%) | n (%) | n (%) |
| Serum Creatinine | Low | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| | High | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Specific Gravity | 1.000 | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| | 1.005 | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| | | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| рН | 5 | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| | 6 | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| | •••• | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Leucocytes | Negative | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| • | Trace | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| | | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Nitrite | Negative | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| | Positive | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Protein (mg/dL) | Negative | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| | Trace | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| | •••• | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Glucose (mg/dL) | Normal | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| | 50 | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| | | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Ketones | Negative | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| | +/small | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| | | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Urobilinogen | Normal | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| | 1 | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| | •••• | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Bilirubin | Negative | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| | + | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| | | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| Blood/Hemoglobin (ery/uL) | Negative | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| | Trace(blood) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |
| | | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) | xx (x.x) |

Table 13: Summary of Anti-tetanus Antibody Titers (IU/mL)

| Visit | Statistics | ITT<br>(N=xx) | Per-protocol<br>(N=xx) |
|---|---|---|---|
| Screening | n | XX | xx |
| | Geometric Mean (SD) | xx.x (x.xx) | xx.x (x.xx) |
| | Min-Max | (xx.x-xx.x) | (xx.x-xx.x) |
| | n | | |
| | Geometric Mean (SD) | xx | |
| Month 1 | Minimum | xx.x (x.xx) | xx |
| | Maximum | XX.X | xx.x (x.xx) |
| | | XX.X | xx.x |
| | | | xx.x |
| (Repeat for all visits) | | | |

Table 14: Summary of Anti-diphtheria Antibody Titers (IU/mL)

| Visit | Statistics | ITT<br>(N=xx) | Per-protocol<br>(N=xx) |
|-----------|---------------------|---------------|------------------------|
| Screening | n | XX | xx |
| | Geometric Mean (SD) | xx.x (x.xx) | xx.x (x.xx) |
| | Min-Max | (xx.x-xx.x) | (xx.x-xx.x) |
| | n | xx | xx |
| Month 1 | Geometric Mean (SD) | xx.x (x.xx) | xx.x (x.xx) |
| | Min-Max | (xx.x-xx.x) | (xx.x-xx.x) |

(Repeat for all visits)

Table 15: Number (%) of Subjects with Post Vaccination Anti-tetanus Antibody Levels

| Visit | Anti-tetanus<br>Antibody Levels | ITT<br>(N=xx) | Per-protocol<br>(N=xx) |
|---|---|---|---|
| Screening | < 5 IU/mL | xx.x (x.xx) | xx.x (x.xx) |
| | ≥ 5 to 10 IU/mL | xx.x (x.xx) | xx.x (x.xx) |
| | ≥10 to 15 IU/mL | xx.x (x.xx) | xx.x (x.xx) |
| | ≥ 15 IU/mL | xx.x (x.xx) | xx.x (x.xx) |
| Month 1 | < 5 IU/mL | xx.x (x.xx) | xx.x (x.xx) |
| | ≥ 5 to 10 IU/mL | xx.x (x.xx) | xx.x (x.xx) |
| | ≥ 10 to 15 IU/mL | xx.x (x.xx) | xx.x (x.xx) |
| | ≥ 15 IU/mL | xx.x (x.xx) | xx.x (x.xx) |

Figure 1: Regression Plot of Reactogenicity versus Anti-diptheria titers - ITT Population



Note: Reactogenicity is defined as the total count of a set of solicited AEs that are expected for up to 3 days after each vaccination.

<sup>&</sup>lt;Program Name: Time and Date>

Figure 2: Plot of GeoMean (± SD) of Tetanus Antibody Titers



Figure 3: Scatter Plot of Percentage of Subjects with Post Vaccination Anti-tetanus Antibody Levels – ITT Population



Figure 4: Scatter Plot of Percentage of Subjects with Post Vaccination Anti-tetanus Antibody Levels – Per-protocol Population



# 14. Appendix B: Listing Shells

| Listing 1. Subject Disposition – Enrolled Subjects | 37 |
|---|---|
| Listing 2. Reasons for Not Meeting Eligibility Criteria – All Subjects | 37 |
| Listing 3. Protocol Deviations – All Subjects | 38 |
| Listing 4. Demographics and Subject Characteristics- ITT Population | 38 |
| Listing 5. Baseline Medical History – ITT Population | 39 |
| Listing 6. Plasmapheresis Check – ITT Population | 39 |
| Listing 7. Previous Immunizations – ITT Population. | 40 |
| Listing 8. Tdap Vaccination – ITT Population | 40 |
| Listing 9. Serum Creatinine and Urinalysis Tests Results – ITT Population | 41 |
| Listing 10. Anti-tetanus and Anti-diptheria Antibody Tests Results – ITT Population | 41 |
| Listing 11. Adverse Events – ITT Population | 42 |
| Listing 12. Solicited Adverse Events – ITT Population | 42 |
| Listing 13. Adverse Events Leading to Withdrawal – ITT Population | 43 |
| Listing 14. Serious Adverse Events – ITT Population | 44 |
| Listing 15. Concomitant Medications – ITT Population | 45 |

Listing 1: Subject Disposition - Enrolled Subjects

| Subject | Consent to | ITT | Per-protocol | Date of Last | Study | Reasons for Early | Reason |
|---|---|---|---|---|---|---|---|
| Number | Study Date | Subject | Subject | Visit/Contact | Completed? | Discontinuation | Detail |
| xxxx | ddmmmyyyy | Y/N | Y/N | ddmmmyyyy | Y/N | xxxxxxx | xxxx |

Programming Note: Subject ID. <pr

Listing 2: Reasons for Not Meeting Eligibility Criteria - All Subjects

| Subject Number | Reason for Screen Failure | Other Description |
|----------------|---------------------------|-------------------|
| xxxx | Subject withdrew consent | |
| | (list all reasons) | |
| | Other: | Verbatim text |

Programming Note: sorted by Subject number.

Listing 3: Protocol Deviations - All Subjects

| Subject<br>Number | <b>Deviation Date</b> | Deviation Detail |
|-------------------|-----------------------|------------------|
| xxxx | dd/mmm/yyyy | Verbatim text |

Note: Only subjects with protocol deviations are listed.

Programming Note: Sorted by Subject number. <Program Name: Time and Date>

Listing 4: Demographics and Subject Characteristics-ITT Population

| Subject | Age at Date of | Gender | Race | Ethnicity |
|---------|-----------------|--------|-------|------------------------|
| Number. | Consent (Years) | | | |
| xxxx | XX | Male | White | Hispanic or Latino |
| | | Female | Other | Not Hispanic of Latino |
| | | | | Not Recorded |

Programming Note: Sorted by subject number. Insert verbatim when "Other" race is selected.

Listing 5: Baseline Medical History - ITT Population

| Subject<br>Number | History<br>Verbatim Term | Start Date | Stop Date | Start Day<br>(relative to start<br>of treatment) | Stop Day<br>(relative to start<br>of treatment) | Ongoing? |
|---|---|---|---|---|---|---|
| xxxx | xxxx | dd/mmm/yyyy | dd/mmm/yyyy | xxx | XXX | Y/N |

Listing 6: Plasmapheresis Check - ITT Population

| Subject Visit | Date of | Eligible for | Inclusion Criteria Not Met |
|---|---|---|---|
| Number | Plasmapheresis Check | Plasmapheresis | |
| xxxx | dd/mmm/yyyy | Yes | Xxxxxxx |

**Listing 7: Previous Immunizations – ITT Population** 

| Subject | Date of Previous | Type of Previous |
|---------|------------------|------------------|
| Number | Immunization | Immunization |
| xxxx | dd/mmm/yyyy | |

Programming Note: Sorted by subject number, exam date.

<Program Name: Time and Date>

Listing 8: Tdap Vaccination - ITT Population

| Subject<br>Number | Date of Tdap<br>Vaccination | Visit | Tdap NDC<br>Number | Tdap Lot<br>Number | Problems with the injection? | Specify |
|---|---|---|---|---|---|---|
| xxxx | dd/mmm/yyyy | Month 0 | | | Y/N | Verbatim text |

Programming Note: Sorted by subject number, exam date.

Listing 9: Serum Creatinine and Urinalysis Tests Results - ITT Population

| Subject<br>Number | Date of<br>Collection | Visit | Test Name (Unit) | Result | Reason not<br>Collected |
|---|---|---|---|---|---|
| xxxx | dd/mmm/yyyy | Screening | Creatinine (Unit) | Xxx | Xxx |
| | | (all Visits) | Glucose | Xxx | Xxx/xx |

Programming Note: Sorted by subject number, Exam Date .

<Program Name: Time and Date>

Listing 10: Anti-tetanus and Anti-diptheria Antibody Tests Results - ITT Population

| Subject<br>Number | Date of<br>Collection | Visit | Plasma Sample<br>Identification # | Test Name (Unit) | Result | Reason not Collected,<br>Specify |
|---|---|---|---|---|---|---|
| xxxx | dd/mmm/yyyy | Screening | | xxx | Xxx | Xxx |
| | | (all Visits) | | xxx/xx | Xxx/xx | Xxx/xx |
| | | Unscheduled | | | | |

Programming Note: Sorted by subject number, Exam Date.

Listing 11: Adverse Events - ITT Population

| Subject<br>Number | AE Name/<br>MedDRA PT <sup>a</sup> /<br>SOC <sup>b</sup> | Onset Date/<br>Stop Date | Onset Day/<br>Duration<br>(Days) | Severity | TEAE/<br>Vaccine<br>Number | Serious?<br>/SAE<br>Description | Outcome | Relationship to<br>Study Product/<br>Action Taken | Other<br>Actions,<br>Specify |
|---|---|---|---|---|---|---|---|---|---|
| xxxx | xxxx/<br>xxxx /<br>xxxx | dd/mmm/yyyy<br>dd/mmm/yyyy<br>or Ongoing | Xx/xx | Mild<br>Moderate<br>Severe | | Y/Xxx<br>N | Resolved<br>Resolved<br>with<br>sequelae | Unrelated<br>Unlikely<br>Possible<br>Probable | |

<sup>a</sup> PT=Preferred Term; <sup>b</sup> SOC=System, Organ, and Class Programming Note: Sorted by Subject Number, Onset Date.

<Program Name: Time and Date>

Listing 12: Solicited Adverse Events - ITT Population

| Subject<br>Number | Vaccination<br>Number | AE Name/<br>MedDRA PT <sup>a</sup> /<br>SOC <sup>b</sup> | Onset Date/<br>Stop Date | Onset Day/<br>Duration<br>(Days) | Severity | TEAE/<br>Vaccine<br>Number | Serious? | Outcome | Relationship to<br>Study Product/<br>Action Taken |
|---|---|---|---|---|---|---|---|---|---|
| xxxx | 1 | xxxx/ | dd/mmm/yyyy | Xx/xx | Mild | | Y | Resolved | Unrelated |
| | 2 | xxxx / | dd/mmm/yyyy | | Moderate | | N | Resolved | Unlikely |
| | | xxxx | or Ongoing | | Severe | | | with<br>sequelae | Possible |
| | | | | | | | | sequerae | Probable |

<sup>a</sup>PT=Preferred Term; <sup>b</sup>SOC=System, Organ, and Class

Note: Solicited AEs reported within the 3 day period after each vaccination is listed.

Programming Note: Sorted by Subject Number, Onset Date.

Listing 13: Adverse Events Leading to Withdrawal – ITT Population

| Subject<br>Number | AE Name/<br>MedDRA PT <sup>a</sup> /<br>SOC <sup>b</sup> | Onset Date/<br>Stop Date | Onset Day/<br>Duration<br>(Days) | Severity | TEAE/<br>Vaccine<br>Number | Serious? | Outcome | Relationship to<br>Study Product/<br>Action Taken | Other<br>Actions,<br>Specify |
|---|---|---|---|---|---|---|---|---|---|
| xxxx | xxxx/<br>xxxx /<br>xxxx | dd/mmm/yyyy<br>dd/mmm/yyyy<br>or Ongoing | Xx/xx | Mild<br>Moderate<br>Severe | | Y/Xxx<br>N | Resolved<br>Resolved<br>with<br>sequelae | Unrelated<br>Unlikely<br>Possible<br>Probable | |

Programming Note: Sorted by Subject Number, Onset Date. <p

a PT=Preferred Term

b SOC=System, Organ, and Class

Listing 14: Serious Adverse Events – ITT Population

| Subject<br>Number | Age (Years)<br>at Screening | Gender | SAE Name | SAE<br>Description | Considered serious because | Onset Date/<br>Stop Date | Vaccination<br>Number | Death Date |
|---|---|---|---|---|---|---|---|---|
| xxxx | xx | Male | Verbatim<br>text | Verbatim<br>text | Death | dd/mmm/yyyy/<br>dd/mmm/yyyy | | dd/mmm/yyyy |
| | | Female | | | Life-threatening | | | |
| | | | | | Hospitalization-initial or<br>prolonged | | | |
| | | | | | Disability or permanent damage | | | |
| | | | | | Congenital anomalies or<br>birth defects | | | |
| | | | | | Other medically important condition | | | |

Programming Note: Sorted by Group, Subject ID. <Program Name: Time and Date>

Listing 14: Serious Adverse Events – ITT Population (continued)

| Subject<br>Number | SAE Name | Hospitalized<br>Date | Discharge<br>Date | Continued Study<br>Participation | Outcome | Relationship to<br>Study Drug | Important<br>Medical Event? |
|---|---|---|---|---|---|---|---|
| xx | Verbatim text | dd/mmm/yyyy | dd/mmm/yyyy | Y/N | Resolved with sequelae | Unrelated<br>Unlikely<br>Possibly Related<br>Probably<br>Related | |
| | | | | | | Definitely<br>Related | |

Programming Note: Sorted by Subject Number. <Program Name: Time and Date>

Listing 15: Concomitant Medications - ITT Population

| Subject<br>Number | Prior<br>Med? | Verbatim<br>Medication Name | Indication | Route | Dose | Frequency | Start Date | Stop Date |
|---|---|---|---|---|---|---|---|---|
| xxx | Y<br>N | xxx | xxxxx | xxxxxx | xxxxxx | xxxxxx | dd/mmm/yyyy | dd/mmm/yyyy<br>or<br>Ongoing |

Programming Note: Sorted by Subject Number, Start Date. <Program Name: Time and Date>